CLINICAL TRIAL: NCT00883181
Title: A Prospective Observational Study of Neutropenia and Anemia Management in Subjects With Solid Tumors Receiving Myelotoxic Chemotherapy
Brief Title: A Study of Neutropenia and Anemia Management in Patients With Solid Tumors Receiving Myelotoxic Chemotherapy
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20060445
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer; Non-Small Cell Lung Cancer; Ovarian Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — This is an observational study. No bio-specimens are being collected.
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective was to describe the incidence of febrile neutropenia based on granulocyte-colony stimulating factor (G-CSF) use (primary, secondary, treatment, or no usage) in patients receiving myelotoxic chemotherapy.

DETAILED DESCRIPTION:
This is a multi-center international observational study of patients receiving myelotoxic regimens, with an investigator assessed risk of febrile neutropenia ≥ 20%, for the treatment of solid tumors (breast, ovarian and lung).

This is an observational study in which patient risk factors were qualitatively (but not quantitatively) assessed, and adherence to G-CSF primary prophylaxis was at the discretion of physicians and not mandated by the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects greater than or equal to 18 years old with breast, ovarian or lung cancer receiving chemotherapy in any schedule, e.g. dose dense or standard chemotherapy.
* These subjects must have an Investigator assessed risk of febrile neutropenia (FN) ≥20% (based on 2006 European Organisation for Research and Treatment of Cancer (EORTC) G-CSF Guidelines

Exclusion Criteria:

- Subjects with concurrent administration of radiotherapy are not eligible (previous radiotherapy is permitted if terminated at least 2 weeks prior to commencing applicable chemotherapy in this study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sites were selected based on where medical data of interest were routinely and completely collected. To avoid geographical bias, sites represented various types of treating centers within each country and sites were encouraged to provide data on patients within all tumor types.
Sampling Method: Probability Sample
Enrollment: 1370 (Actual)
Dates: Start 2006-11; Primary Completion 2009-10 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Maenpaa J, Varthalitis I, Erdkamp F, Trojan A, Krzemieniecki K, Lindman H, Bendall K, Vogl FD, Verma S. The use of granulocyte colony stimulating factor (G-CSF) and management of chemotherapy delivery during adjuvant treatment for early-stage breast cancer--further observations from the IMPACT solid study. Breast. 2016 Feb;25:27-33. doi: 10.1016/j.breast.2015.11.007. Epub 2015 Dec 20. PMID 26801413
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1370 patients were enrolled at 87 sites in Europe, 5 sites in Canada, and 10 sites in Australia from December 2007 to October 2009. Of these, 1347 participants were included in the full analysis set (FAS) consisting of all enrolled patients who met protocol defined eligibility criteria and started at least 1 cycle of chemotherapy.
Pre-assignment Details: Eligible patients were enrolled sequentially. Upon completion of all planned chemotherapy cycles, or following cessation of chemotherapy for any reason, patients were followed-up annually for 5 years or until disease progression or death.
Groups:
- Full Analysis Set: Participants diagnosed with breast, ovarian, or lung cancer and receiving myelotoxic chemotherapy.
Period: Overall Study
Arm/Group | Full Analysis Set
Started | 1347 (Full analysis set)
Completed | 1069 (Completed planned chemotherapy)
Not Completed | 278
Not completed — Hematological Adverse Event | 26
Not completed — Non-hematological Adverse Event | 55
Not completed — Disease Progression | 94
Not completed — Administrative Reason | 24
Not completed — Withdrawal by Subject | 4
Not completed — Death | 31
Not completed — Other | 38
Not completed — Protocol Deviation | 3
Not completed — Noncompliance | 3

BASELINE CHARACTERISTICS:
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 1347
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1072
  Male | 275
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 1324
  Black or African American | 4
  Hispanic or Latino | 3
  Asian | 4
  Other | 4
  Not Applicable | 8
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature; 2 = Ambulatory and capable of all self care, unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    0 - Normal Activity | 874
    1 - Symptoms but Ambulatory | 346
    2 - Confined to Bed ≤ 50% of Time | 99
    3 - Confined to Bed ≥ 50% of Time | 9
    4 - 100% Bedridden | 0
    Missing | 19
Tumor Type [Number; unit: participants]
  Ovarian cancer | 157
  Non-small cell lung cancer (NSCLC) | 224
  Small cell lung cancer (SCLC) | 137
  Breast cancer | 829
Prior Treatment [Number; unit: participants]
  None | 647
  Chemotherapy only | 88
  Radiotherapy only | 19
  Chemotherapy and radiotherapy | 62
  Surgery | 449
  Other | 80
  Missing | 2
Prior Febrile Neutropenia Episodes [Number; unit: participants] — Episodes of febrile neutropenia (FN) that occurred during prior cancer treatment; 698 participants had received prior treatment.
  participants
    Any prior FN episodes | 35
    No prior FN episodes | 213
    Missing | 450
Hemoglobin Level [Number; unit: participants]
  < 11 g/dL | 175
  ≥ 11 g/dL | 1091
  Missing | 81
Anemia Symptoms [Number; unit: participants] — Anemia symptoms were available for 692 participants at baseline. Participants may have more than one anemia symptom.
  participants
    Fatigue/tiredness | 197
    Pallor/Pale skin | 86
    Headache | 53
    Dyspnea | 101
    Tachycardia and/or palpitations | 48
    Dizziness and/or vertigo | 49
    Irritability | 66
    Depression | 113
    Nausea | 38
    Anorexia | 65
    Impaired cognitive function | 17
    Impaired immune system | 12
    Metabolic dysfunction | 32
    Sexual dysfunction | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Febrile Neutropenia (FN)
Description: Febrile neutropenia was defined as a single oral temperature ≥ 38.3°C, or a temperature of ≥ 38.0°C for ≥ 1 hour with a neutrophil count of < 500 cells/mm² or < 1000 cells/mm² and predicted to fall below 500 cells/mm².
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set; Note: One participant with breast cancer had disease stage missing.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ovarian: Participants diagnosed with ovarian cancer and receiving chemotherapy.
- NSCLC: Participants diagnosed with non-small cell lung cancer (NSCLC) and receiving chemotherapy.
- SCLC: Participants diagnosed with small cell lung cancer (SCLC) and receiving chemotherapy.
- Breast Stage I-III: Participants diagnosed with Stage I-III breast cancer and receiving chemotherapy.
- Breast Metastatic: Participants diagnosed with metastatic breast cancer and receiving chemotherapy.
- Breast Total: Participants diagnosed with breast cancer (any stage) and receiving chemotherapy.
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 157 | 224 | 137 | 738 | 90 | 829
percentage of participants | 8 [4 to 13] | 8 [5 to 12] | 15 [10 to 21] | 9 [7 to 11] | 11 [6 to 19] | 9 [7 to 11]

2. Secondary Outcome: Number of Participants Who Received G-CSF During Cycles 1 to 8
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 157 | 224 | 137 | 738 | 90 | 829
participants
  Primary Prophylaxis - Pegfilgrastim | 24 | 22 | 33 | 360 | 32 | 393
  Primary Prophylaxis - Any Daily G-CSF | 6 | 20 | 11 | 51 | 6 | 57
  Primary Prophylaxis - Other G-CSF | 1 | 3 | 0 | 6 | 1 | 7
  Secondary Prophylaxis - Pegfilgrastim | 11 | 14 | 15 | 92 | 9 | 101
  Secondary Prophylaxis - Any Daily G-CSF | 15 | 24 | 13 | 64 | 9 | 73
  Secondary Prophylaxis - Other G-CSF | 4 | 3 | 0 | 1 | 1 | 2
  Treatment - Pegfilgrastim | 5 | 2 | 1 | 0 | 0 | 0
  Treatment - Any Daily G-CSF | 9 | 15 | 8 | 17 | 4 | 21
  Treatment - Other G-CSF | 0 | 1 | 0 | 0 | 0 | 0
  No G-CSF Used | 82 | 120 | 56 | 147 | 28 | 175

3. Primary Outcome: Percentage of Participants Who Received No Prophylaxis or Treatment With Granulocyte Colony-stimulating Factors (G-CSF) Who Experienced Febrile Neutropenia
Description: FN was defined as a single oral temperature ≥ 38.3°C, or a temperature of ≥ 38.0°C for ≥ 1 hour with a neutrophil count of < 500 cells/mm² or < 1000 cells/mm² and predicted to fall below 500 cells/mm². Assignment to G-CSF use groups was programmatically derived rather than assigned by the investigator. Participants in the No G-CSF use group received no G-CSF prophylaxis or treatment at any time during cycles 1 to 8.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received no prophylaxis or treatment with any G-CSF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 82 | 120 | 56 | 147 | 28 | 175
percentage of participants | 4 [1 to 10] | 3 [1 to 7] | 5 [2 to 15] | 1 [1 to 4] | 0 [NA to NA] — Not calculated when n=0 | 1 [1 to 3]

4. Primary Outcome: Percentage of Participants Receiving Primary Prophylaxis With Pegfilgrastim Who Experienced Febrile Neutropenia
Description: FN was defined as a single oral temperature ≥ 38.3°C, or a temperature of ≥ 38.0°C for ≥ 1 hour with a neutrophil count of < 500 cells/mm² or < 1000 cells/mm² and predicted to fall below 500 cells/mm². Primary prophylaxis with pegfilgrastim was defined as receiving pegfilgrastim starting in cycle 1 on day 1 to 7 if chemotherapy completed by day 7 and day 1 to 11 if chemotherapy completed after day 7. Assignment to G-CSF use groups was programmatically derived rather than assigned by the investigator. Participants were assigned to a G-CSF use group that represented the 'best' G-CSF therapy they received at any point in the study. Participants who received G-CSF support from the beginning of Cycle 1 were assigned to primary prophylaxis regardless of whether they continued to receive G-CSF support in subsequent cycles.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received primary prophylaxis with pegfilgrastim
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 24 | 22 | 33 | 360 | 32 | 393
percentage of participants | 0 [NA to NA] — Not calculated when n=0 | 0 [NA to NA] — Not calculated when n=0 | 21 [11 to 38] | 9 [7 to 13] | 9 [3 to 24] | 9 [7 to 13]

5. Primary Outcome: Percentage of Participants Receiving Primary Prophylaxis With Any Daily G-CSF Who Experienced Febrile Neutropenia
Description: FN was defined as a single oral temperature ≥ 38.3°C, or a temperature of ≥ 38.0°C for ≥ 1 hour with a neutrophil count of < 500 cells/mm² or < 1000 cells/mm² and predicted to fall below 500 cells/mm². Primary prophylaxis was defined as receiving any daily G-CSF (e.g. filgrastim or lenograstim) starting in cycle 1 on day 1 to 7 if chemotherapy completed by day 7 and day 1 to 11 if chemotherapy completed after day 7. Assignment to G-CSF use groups was programmatically derived rather than assigned by the investigator. Participants were assigned to a G-CSF use group that represented the 'best' G-CSF therapy they received at any point in the study. Participants who received G-CSF support from the beginning of cycle 1 were assigned to primary prophylaxis regardless of whether they continued to receive G-CSF support in subsequent cycles.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received primary prophylaxis with any daily G-CSF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 6 | 20 | 11 | 51 | 6 | 57
percentage of participants | 0 [NA to NA] — Not calculated when n=0 | 20 [8 to 42] | 9 [2 to 38] | 6 [2 to 16] | 17 [3 to 56] | 7 [3 to 17]

6. Primary Outcome: Percentage of Participants Receiving Secondary Prophylaxis With Pegfilgrastim Who Experienced Febrile Neutropenia
Description: FN was defined as a single oral temperature ≥ 38.3°C, or a temperature of ≥ 38.0°C for ≥ 1 hour with a neutrophil count of < 500 cells/mm² or < 1000 cells/mm² and predicted to fall below 500 cells/mm². Secondary prophylaxis with pegfilgrastim was defined as receiving pegfilgrastim starting in cycle 2 onwards on day 1 to 7 if chemotherapy completed by day 7 and day 1 to 11 if chemotherapy completed after day 7. Assignment to G-CSF use groups was programmatically derived rather than assigned by the investigator. Participants were assigned to a G-CSF use group that represented the 'best' G-CSF therapy they received at any point in the study. Adherence of G-CSF support in subsequent cycles was not required for secondary prophylaxis; just an initiation of pegfilgrastim support in the beginning of cycle 2 or later. Results include the FN event that may have triggered the secondary prophylaxis treatment.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received secondary prophylaxis with pegfilgrastim
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 11 | 14 | 15 | 92 | 9 | 101
percentage of participants | 0 [NA to NA] — Not calculated when n=0 | 36 [16 to 61] | 40 [20 to 64] | 14 [8 to 23] | 33 [12 to 65] | 16 [10 to 24]

7. Primary Outcome: Percentage of Participants Receiving Secondary Prophylaxis With Any Daily G-CSF Who Experienced Febrile Neutropenia
Description: FN was defined as a single oral temperature ≥ 38.3°C, or a temperature of ≥ 38.0°C for ≥ 1 hour with a neutrophil count of < 500 cells/mm² or < 1000 cells/mm² and predicted to fall below 500 cells/mm². Secondary prophylaxis was defined as receiving any daily G-CSF starting in cycle 2 onwards on day 1 to 7 if chemotherapy completed by day 7 and day 1 to 11 if chemotherapy completed after day 7. Assignment to G-CSF use groups was programmatically derived rather than assigned by the investigator. Participants were assigned to a G-CSF use group that represented the 'best' G-CSF therapy they received at any point in the study. Adherence of G-CSF support in subsequent cycles was not required for secondary prophylaxis; just an initiation of G-CSF support in the beginning of cycle 2 or later. Results include the FN event that may have triggered the secondary prophylaxis treatment.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received secondary prophylaxis with any daily G-CSF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 15 | 24 | 13 | 64 | 9 | 73
percentage of participants | 27 [11 to 52] | 13 [4 to 31] | 15 [4 to 42] | 20 [12 to 32] | 22 [6 to 55] | 21 [13 to 31]

8. Secondary Outcome: Number of Days of Prophylaxis in Participants Receiving Primary Prophylaxis With Pegfilgrastim
Description: The average number of days of pegfilgrastim use per cycle was calculated across all administered cycles.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received primary prophylaxis with pegfilgrastim
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 24 | 22 | 33 | 360 | 32 | 393
days | 1.00 (0.00) [NA to NA] | 1.00 (0.00) [NA to NA] | 1.01 (0.03) [11 to 38] | 1.00 (0.05) [7 to 13] | 1.01 (0.03) [3 to 24] | 1.00 (0.04) [7 to 13]

9. Secondary Outcome: Number of Days of Prophylaxis in Participants Receiving Primary Prophylaxis With Any Daily G-CSF
Description: The average number of days of daily G-CSF use per cycle was calculated across all administered cycles.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received primary prophylaxis with any daily G-CSF
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 6 | 20 | 11 | 51 | 6 | 57
days | 3.67 (1.63) [NA to NA] | 3.95 (1.18) [8 to 42] | 4.95 (1.31) [2 to 38] | 4.77 (1.72) [2 to 16] | 5.85 (2.64) [3 to 56] | 4.88 (1.84) [3 to 17]

10. Secondary Outcome: Number of Days of Prophylaxis in Participants Receiving Secondary Prophylaxis With Pegfilgrastim
Description: The average number of days of pegfilgrastim use per cycle was calculated across all administered cycles.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received secondary prophylaxis with pegfilgrastim
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 11 | 14 | 15 | 92 | 9 | 101
days | 1.00 (0.00) [NA to NA] | 1.00 (0.00) [16 to 61] | 1.04 (0.12) [20 to 64] | 1.02 (0.21) [8 to 23] | 1.00 (0.00) [12 to 65] | 1.02 (0.20) [10 to 24]

11. Secondary Outcome: Number of Days of Prophylaxis in Participants Receiving Secondary Prophylaxis With Any Daily G-CSF
Description: The average number of days of daily G-CSF use per cycle was calculated across all administered cycles.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received secondary prophylaxis with any daily G-CSF.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 15 | 24 | 13 | 64 | 9 | 73
days | 3.66 (1.82) [11 to 52] | 4.28 (0.87) [4 to 31] | 4.04 (1.61) [4 to 42] | 4.74 (2.64) [12 to 32] | 3.50 (0.95) [6 to 55] | 4.58 (2.53) [13 to 31]

12. Primary Outcome: Percentage of Participants Receiving Primary Prophylaxis With an Other G-CSF Who Experienced Febrile Neutropenia
Description: FN was defined as a single oral temperature ≥ 38.3°C, or a temperature of ≥ 38.0°C for ≥ 1 hour with a neutrophil count of < 500 cells/mm² or < 1000 cells/mm² and predicted to fall below 500 cells/mm². Primary prophylaxis was defined as receiving any other G-CSF starting in cycle 1 on day 1 to 7 if chemotherapy completed by day 7 and day 1 to 11 if chemotherapy completed after day 7. Assignment to G-CSF use groups was programmatically derived rather than assigned by the investigator. Participants were assigned to a G-CSF use group that represented the 'best' G-CSF therapy they received at any point in the study. Participants who received G-CSF support from the beginning of cycle 1 were assigned to primary prophylaxis regardless of whether they continued to receive G-CSF support in subsequent cycles.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received primary prophylaxis with other G-CSF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 1 | 3 | 0 | 6 | 1 | 7
percentage of participants | 0 [NA to NA] — Not calculated when n=0 | 0 [NA to NA] — Not calculated when n=0 |  | 17 [3 to 56] | 0 [NA to NA] — Not calculated when n=0 | 14 [3 to 51]

13. Primary Outcome: Percentage of Participants Receiving Secondary Prophylaxis With an Other G-CSF Who Experienced Febrile Neutropenia
Description: as for outcome 7
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received secondary prophylaxis with other G-CSF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 4 | 3 | 0 | 1 | 1 | 2
percentage of participants | 25 [5 to 70] | 0 [NA to NA] — Not calculated when n=0 |  | 0 [NA to NA] — Not calculated when n=0 | 0 [NA to NA] — Not calculated when n=0 | 0 [NA to NA] — Not calculated when n=0

14. Primary Outcome: Percentage of Participants Receiving Treatment With Pegfilgrastim Who Experienced Febrile Neutropenia
Description: FN was defined as a single oral temperature ≥ 38.3°C, or a temperature of ≥ 38.0°C for ≥ 1 hour with a neutrophil count of < 500 cells/mm² or < 1000 cells/mm² and predicted to fall below 500 cells/mm². Treatment with pegfilgrastim is defined as participants who started pegfilgrastim treatment after day 7 of any cycle if chemotherapy completed by day 7 and after day 11 of any cycle if chemotherapy completed after day 7.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received treatment with pegfilgrastim
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 5 | 2 | 1 | 0 | 0 | 0
percentage of participants | 0 [NA to NA] — Not calculated when n=0 | 0 [NA to NA] — Not calculated when n=0 | 0 [NA to NA] — Not calculated when n=0 |  |  |

15. Primary Outcome: Percentage of Participants Receiving Treatment With Any Daily G-CSF Who Experienced Febrile Neutropenia
Description: FN was defined as a single oral temperature ≥ 38.3°C, or a temperature of ≥ 38.0°C for ≥ 1 hour with a neutrophil count of < 500 cells/mm² or < 1000 cells/mm² and predicted to fall below 500 cells/mm². Treatment with any daily G-CSF is defined as participants who started daily G-CSF treatment after day 7 of any cycle if chemotherapy completed by day 7 and after day 11 of any cycle if chemotherapy completed after day 7.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received treatment with any daily G-CSF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 9 | 15 | 8 | 17 | 4 | 21
percentage of participants | 44 [19 to 73] | 13 [4 to 38] | 13 [2 to 47] | 12 [3 to 34] | 25 [5 to 70] | 14 [5 to 35]

16. Primary Outcome: Percentage of Participants Receiving Treatment With Any Other G-CSF Who Experienced Febrile Neutropenia
Description: FN was defined as a single oral temperature ≥ 38.3°C, or a temperature of ≥ 38.0°C for ≥ 1 hour with a neutrophil count of < 500 cells/mm² or < 1000 cells/mm² and predicted to fall below 500 cells/mm². Treatment with any other G-CSF is defined as participants who started other G-CSF treatment after day 7 of any cycle if chemotherapy completed by day 7 and after day 11 of any cycle if chemotherapy completed after day 7.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received treatment with any other G-CSF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
percentage of participants |  | 100 [NA to NA] — Not calculated when n=100 |  |  |  |

17. Secondary Outcome: Number of Days of Treatment in Participants Receiving Treatment With Pegfilgrastim
Description: The average number of days of pegfilgrastim use per cycle was calculated across all administered cycles.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received treatment with pegfilgrastim
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 5 | 2 | 1 | 0 | 0 | 0
days | 1.40 (0.89) | 1.00 (0.00) | 1.00 (NA) — Not calculated as N=1 |  |  |

18. Secondary Outcome: Number of Days of Treatment in Participants Receiving Treatment With Any Daily G-CSF
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants who received treatment with any daily G-CSF
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 9 | 15 | 8 | 17 | 4 | 21
days | 3.11 (1.92) [19 to 73] | 4.45 (1.18) [4 to 38] | 2.83 (1.21) [2 to 47] | 2.95 (1.50) [3 to 34] | 2.38 (0.75) [5 to 70] | 2.84 (1.39) [5 to 35]

19. Secondary Outcome: Percentage of Participants With Chemotherapy Dose Delays in Cycles 2 Through 8
Description: A dose delay is defined as a delay of more than 3 days in the start of chemotherapy measured since the start of the previous cycle. The percentage of participants with delays in chemotherapy administration are summarized by the length of delay (> 3 days, > 5 days, and > 7 days) across cycles 2 through 8.
Time Frame: Cycles 2 - 8 (approximately 21 weeks)
Population: Full analysis set participants who received more than 1 cycle of chemotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 147 | 204 | 124 | 734 | 87 | 822
percentage of participants
  > 3 Days Delay in One or More Cycles | 48 [40 to 56] | 46 [39 to 52] | 52 [44 to 61] | 29 [26 to 32] | 47 [37 to 58] | 31 [28 to 34]
  > 5 Days Delay in One or More Cycles | 39 [32 to 48] | 39 [33 to 46] | 47 [38 to 56] | 22 [19 to 25] | 40 [31 to 51] | 24 [21 to 27]
  > 7 Days Delay in One or More Cycles | 24 [18 to 31] | 23 [18 to 29] | 26 [19 to 34] | 9 [7 to 11] | 21 [14 to 30] | 10 [8 to 12]

20. Secondary Outcome: Percentage of Cycles With Chemotherapy Dose Delays
Description: A dose delay is defined as a delay of > 3 days in the start of chemotherapy measured since the start of the previous cycle. The percentage of cycles delayed are summarized by the length of delay (> 3 days, > 5 days, and > 7 days) across cycles 2 through 8.
Time Frame: Cycles 2 - 8 (approximately 21 days)
Population: Full analysis set participants who received more than 1 cycle of chemotherapy
Measure: Number; unit: percentage of cycles
Units Other Than Participants: Total cycles
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 147 | 204 | 124 | 734 | 87 | 822
Number analyzed (Total cycles) | 622 | 585 | 473 | 3697 | 402 | 4104
percentage of cycles
  > 3 Days Delay in One or More Cycles | 20 | 24 | 24 | 7 | 17 | 8
  > 5 Days Delay in One or More Cycles | 16 | 19 | 19 | 5 | 14 | 6
  > 7 Days Delay in One or More Cycles | 7 | 9 | 8 | 2 | 6 | 2 [upper limit 12]

21. Secondary Outcome: Percentage of Participants With Chemotherapy Dose Reductions
Description: A participant is considered to have a dose reduction in a given cycle if there was a ≥ 15% reduction in dose of any chemotherapy agent planned for that cycle, relative to the dose planned at the baseline visit for that cycle.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants with actual regimens as planned (17 participants received a different regimen to what was planned and are thus excluded)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 152 | 219 | 137 | 732 | 89 | 822
percentage of participants | 34 [27 to 42] | 25 [20 to 31] | 22 [16 to 30] | 16 [13 to 19] | 29 [21 to 39] | 17 [15 to 20]

22. Secondary Outcome: Percentage of Cycles With Chemotherapy Dose Reductions
Description: A dose reduction in a given cycle is defined as a ≥ 15% reduction in dose of any chemotherapy agent planned for that cycle, relative to the dose planned at the baseline visit for that cycle.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: as for outcome 21
Measure: Number; unit: percentage of cycles
Units Other Than Participants: Total cycles
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 152 | 219 | 137 | 732 | 89 | 822
Number analyzed (Total cycles) | 757 | 791 | 610 | 4399 | 486 | 4891
percentage of cycles | 16 [27 to 42] | 13 [20 to 31] | 12 [16 to 30] | 6 [13 to 19] | 16 [21 to 39] | 7 [15 to 20]

23. Secondary Outcome: Reasons for Cycles With > 3 Days Chemotherapy Dose Delays in Cycles 2 to 8
Description: A dose delay is defined as a delay of > 3 days in the start of chemotherapy measured since the start of the previous cycle.
Time Frame: Cycles 2 - 8 (approximately 21 weeks)
Population: Full analysis set participants who received more than 1 cycle of chemotherapy and had > 3 days delay in one or more cycles
Measure: Number; unit: cycles
Units Other Than Participants: Cycles with > 3 days delay
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 71 | 93 | 65 | 212 | 41 | 253
Number analyzed (Cycles with > 3 days delay) | 124 | 142 | 113 | 268 | 70 | 338
cycles
  Febrile Neutropenia | 1 | 6 | 6 | 12 | 3 | 15
  Chemotherapy Induced Neutropenia | 27 | 34 | 14 | 41 | 9 | 50
  Chemotherapy Induced Anemia | 5 | 7 | 1 | 3 | 0 | 3 [upper limit 12]
  Chemotherapy Induced Thrombocytopenia | 7 | 0 | 4 | 1 | 1 | 2
  Other Hematological Reason | 2 | 1 | 1 | 8 | 2 | 10
  Gastrointestinal Toxicity | 3 | 0 | 2 | 3 | 1 | 4
  Neurological Toxicity | 3 | 2 | 1 | 5 | 3 | 8
  Hepatic Toxicity | 1 | 0 | 1 | 4 | 0 | 4
  Other Non-Hematological Reason | 14 | 21 | 20 | 44 | 6 | 50
  Dose Administration Error | 0 | 3 | 0 | 0 | 0 | 0
  Participant Preference | 19 | 19 | 15 | 51 | 16 | 67
  Other | 24 | 33 | 34 | 78 | 19 | 97
  Missing | 18 | 16 | 14 | 18 | 10 | 28

24. Secondary Outcome: Reasons for Cycles With ≥ 15% Chemotherapy Dose Reductions in Cycles 1-8
Description: as for outcome 22
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set participants with actual regimens as planned and with ≥ 15% chemotherapy dose reduction in any cycle.
Measure: Number; unit: cycles
Units Other Than Participants: Cycles with ≥ 15% dose reduction
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 52 | 55 | 30 | 116 | 26 | 142
Number analyzed (Cycles with ≥ 15% dose reduction) | 123 | 99 | 71 | 256 | 77 | 333
cycles
  Febrile neutropenia | 4 [27 to 42] | 4 [20 to 31] | 3 [16 to 30] | 15 [13 to 19] | 6 [21 to 39] | 21 [15 to 20]
  Chemotherapy induced neutropenia | 15 | 16 | 3 | 41 | 11 | 52
  Chemotherapy induced anemia | 3 | 7 | 2 | 2 | 0 | 2
  Chemotherapy induced thrombocytopenia | 5 | 4 | 2 | 0 | 1 | 1
  Other hematological reason | 1 | 1 | 2 | 0 | 0 | 0
  Gastrointestinal toxicity | 4 | 2 | 1 | 12 | 2 | 14
  Neurological toxicity | 2 | 2 | 2 | 17 | 0 | 17
  Hepatic toxicity | 0 | 1 | 2 | 0 | 0 | 0
  Other non-hematological reason | 31 | 13 | 10 | 33 | 8 | 41
  Weight loss | 1 | 1 | 5 | 0 | 1 | 1
  Dose administration error | 1 | 0 | 0 | 1 | 2 | 3
  Participant preference | 2 | 0 | 0 | 0 | 0 | 0
  Reduced to assess dose/tolerability | 2 | 6 | 1 | 6 | 1 | 7
  Other | 16 | 19 | 11 | 20 | 10 | 30
  Missing | 36 | 23 | 27 | 109 | 35 | 144

25. Secondary Outcome: Number of Participants With Systemic Anti-infective Use in Cycles 1 to 8
Description: Number of participants with systemic anti-infective use, including antibiotics, anti-fungal and virostatic for prophylaxis or treatment.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 157 | 224 | 137 | 738 | 90 | 829
participants | 23 | 46 | 53 | 198 | 20 | 218

26. Secondary Outcome: Number of Participants With Unplanned Hospitalizations
Description: Unplanned hospitalizations included only those which involved an overnight stay and occurred in cycles 1 to 8.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 157 | 224 | 137 | 738 | 90 | 829
participants | 26 | 52 | 41 | 107 | 18 | 125

27. Secondary Outcome: Investigator Assessed Clinical Response at End of Treatment
Time Frame: End of treatment (approximately 24 weeks)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 157 | 224 | 137 | 738 | 90 | 829
participants
  Complete response | 49 | 8 | 17 | 218 | 4 | 222
  Partial response | 29 | 60 | 38 | 77 | 36 | 114
  Stable disease/No response | 23 | 41 | 29 | 35 | 11 | 46
  Progressive disease | 31 | 64 | 33 | 8 | 18 | 26
  Not done | 25 | 51 | 20 | 383 | 21 | 404
  Missing | 0 | 0 | 0 | 17 | 0 | 17

28. Secondary Outcome: Number of Participants With Hematological Toxicities
Description: The number of participants experiencing treatment related grade 3 and 4 hematological toxicities during cycles 1 to 8. Participants experiencing both Grade 3 and Grade 4 toxicities are reported under Grade 4 only (maximum toxicity). Toxicity grades for hematology data are defined according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0: Absolute neutrophil count (ANC) - Grade 3: < 1.0 - 0.5 x 10^9/L; ANC - Grade 4: < 0.5 x 10^9/L; White blood cells (WBC) - Grade 3: < 2.0 - 1.0 x 10^9/L; WBC - Grade 4: < 1.0 x 10^9/L; Hemoglobin - Grade 3: < 8.0 - 6.5 g/dL; Hemoglobin - Grade 4: < 6.5 g/dL; Platelets - Grade 3: < 50 - 25 x 10^9/L; Platelets - Grade 4: < 25 x 10^9/L.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 157 | 224 | 137 | 738 | 90 | 829
participants
  Grade 3 absolute neutrophil count | 19 | 7 | 9 | 45 | 5 | 50
  Grade 4 absolute neutrophil count | 23 | 18 | 13 | 89 | 18 | 107
  Grade 3 white blood cells | 17 | 11 | 5 | 71 | 8 | 79
  Grade 4 white blood cells | 6 | 8 | 11 | 38 | 12 | 50
  Grade 3 hemoglobin | 6 | 12 | 15 | 47 | 7 | 54
  Grade 4 hemoglobin | 1 | 6 | 5 | 9 | 3 | 12
  Grade 3 platelets | 8 | 2 | 3 | 6 | 3 | 9
  Grade 4 platelets | 3 | 3 | 4 | 3 | 0 | 3

29. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was calculated from cycle 1 day 1 to a date at which disease progression was first recorded. Participants who died due to causes other than disease progression were censored at the date of death. Participants who were alive and whose disease had not progressed at the most recent contact, or who were lost to follow-up, or with missing data, were censored at the date of last contact. Median time to disease progression was estimated from the Kaplan-Meier survival function.
Time Frame: From cycle 1, day 1 until end of the long-term follow-up; median time on follow-up from cycle 1, day 1 was 52 months.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 157 | 224 | 137 | 738 | 90 | 829
months | 12.4 [9.9 to 16.4] | 6.5 [4.5 to 7.8] | 6.8 [6.4 to 7.9] | NA [NA to NA] — Not estimable due to the low number of events | 11.8 [9.1 to 16.4] | NA [NA to NA] — Not estimable due to the low number of events

30. Secondary Outcome: Duration of Treatment With Erythropoiesis-stimulating Agents (ESAs)
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Participants who received treatment with an ESA
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 147
weeks | 5.3 (4.6)

31. Secondary Outcome: Reason for Treatment With Erythropoiesis-stimulating Agents
Description: The reason treatment with an ESA was initiated as recorded by the investigator; participants may have more than one reason for initiating treatment.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Participants who received treatment with an ESA
Measure: Number; unit: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 147
participants
  Hemoglobin level | 134 (4.6)
  Risk of chemotherapy induced anemia | 10
  Evidence based guidelines | 3
  Other anemia-related symptoms | 3

32. Secondary Outcome: Hemoglobin Level at Initiation of Erythropoiesis-stimulating Agent Treatment
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Participants who received treatment with an ESA
Measure: Number; unit: participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 147
participants
  Hemoglobin < 9 g/dL | 19 (4.6)
  Hemoglobin 9 - 11 g/dL | 95
  Hemoglobin > 11 g/dL | 29
  Missing | 4

33. Secondary Outcome: Number of Clinical Visits in Cycles 1-8 by ESA Use
Description: The average number of clinical visits per month (28 day period) during cycles 1 to 8 and during the period of ESA treatment in cycles 1 to 8.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: visits per month
Groups:
- Any ESA Use: Participants who received treatment with any erythropoiesis-stimulating agent (ESA) during cycles 1 to 8.
- No ESA Use: Participants who did not receive treatment with a erythropoiesis-stimulating agent (ESA) during cycles 1 to 8.
Arm/Group | Any ESA Use | No ESA Use
Number analyzed (Participants) | 147 | 1200
visits per month
  Visits per month during cycles 1 - 8 | 3.1 (1.6) | 2.8 (1.7)
  Visits per month during period of ESA treatment | 3.9 (3.2) | NA (NA) — Participants in this group did not receive any ESA treatment

34. Secondary Outcome: Percentage of Participants Who Received ESAs and Required a Red Blood Cell (RBC) Transfusion After 5 Weeks of ESA Treatment
Description: Kaplan-Meier estimate of the percentage of participants with RBC transfusions from five weeks post initiation of ESA treatment until the end of ESA treatment during cycles 1 to 8.
Time Frame: From 5 weeks post initiation of ESA treatment to the end of ESA treatment phase (EOTP) during cycles 1 - 8; maximum duration of ESA treatment was 23 weeks.
Population: Participants who received treatment with an ESA and still on study 5 weeks after initiation of ESA treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 105
percentage of participants | 11 (4.6) [3 to 19]

35. Secondary Outcome: Change in Hemoglobin During ESA Treatment Phase
Time Frame: Initiation of ESA treatment (last assessment on or prior to ESA day 1) and at end of ESA treatment; median duration of ESA treatment was 4 weeks, maximum was 23 weeks.
Population: Participants who received treatment with an ESA and with hemoglobin measurements available at both time points.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 121
g/dL | 0.38 (1.30)

36. Secondary Outcome: Percentage of Participants Who Received ESAs and Achieved Hematopoietic Response
Description: Kaplan-Meier estimate of the percentage of participants in cycles 1 to 8 receiving ESA treatment who achieved a hematopoietic response during the ESA treatment phase, defined as a hemoglobin concentration ≥ 12 g/dL or a ≥ 2 g/dL rise in hemoglobin after starting ESA treatment.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Participants who received treatment with an ESA
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 147
percentage of participants | 45 (4.6) [29 to 61]

37. Secondary Outcome: Percentage of Participants Who Received ESAs and Achieved Hemoglobin ≥ 9 g/dL After 5 Weeks ESA Treatment
Description: Kaplan-Meier estimate of the percentage of participants achieving a hemoglobin level ≥ 9 g/dL during the period from five weeks after initiation of ESA treatment until the end of ESA treatment during cycles 1 to 8.
Time Frame: as for outcome 34
Population: Participants who received treatment with an ESA and with hemoglobin < 9 g/dL at initiation of ESA treatment and still on study 5 weeks after initiation of ESA treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 14
percentage of participants | 58 (4.6) [-1 to 118]

38. Secondary Outcome: Percentage of Participants Who Received ESAs and Achieved Hemoglobin ≥ 10 g/dL After 5 Weeks ESA Treatment
Description: Kaplan-Meier estimate of the percentage of participants achieving a hemoglobin level ≥ 10 g/dL during the period from five weeks after initiation of ESA treatment until the end of ESA treatment during cycles 1 to 8.
Time Frame: as for outcome 34
Population: Participants who received treatment with an ESA, and with hemoglobin < 10 g/dL at initiation of ESA treatment and still on study 5 weeks after initiation of ESA treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 41
percentage of participants | 85 (4.6) [61 to 108]

39. Secondary Outcome: Percentage of Participants Who Received ESAs and Achieved Hemoglobin ≥ 11 g/dL After 5 Weeks ESA Treatment
Description: Kaplan-Meier estimate of the percentage of participants achieving a hemoglobin level ≥ 11 g/dL during the period from five weeks after initiation of ESA treatment until the end of ESA treatment during cycles 1 to 8.
Time Frame: as for outcome 34
Population: Participants who received treatment with an ESA, and with hemoglobin < 11 g/dL at initiation of ESA treatment and still on study 5 weeks after initiation of ESA treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 82
percentage of participants | 66 (4.6) [51 to 82]

40. Secondary Outcome: Percentage of Participants Who Received ESAs and Achieved Hemoglobin ≥ 12 g/dL After 5 Weeks ESA Treatment
Description: Kaplan-Meier estimate of the percentage of participants achieving a hemoglobin level ≥ 12 g/dL during the period from five weeks after initiation of ESA treatment until the end of ESA treatment during cycles 1 to 8.
Time Frame: as for outcome 34
Population: Participants who received treatment with an ESA, and with hemoglobin < 12 g/dL at initiation of ESA treatment and still on study 5 weeks after initiation of ESA treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 97
percentage of participants | 35 (4.6) [17 to 53]

41. Secondary Outcome: Percentage of Participants Who Received ESAs and Achieved Hemoglobin From 10 to 12 g/dL After 5 Weeks ESA Treatment
Description: Kaplan-Meier estimate of the percentage of participants achieving a hemoglobin level from 10 to 12 g/dL during the period from five weeks after initiation of ESA treatment until the end of ESA treatment during cycles 1 to 8.
Time Frame: as for outcome 34
Population: as for outcome 38
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 41
percentage of participants | 84 (4.6) [58 to 109]

42. Secondary Outcome: Percentage of Participants Who Received ESAs and Achieved Hemoglobin From 12 to 13 g/dL After 5 Weeks ESA Treatment
Description: Kaplan-Meier estimate of the percentage of participants achieving a hemoglobin level from 12 to 13 g/dL during the period from five weeks after initiation of ESA treatment until the end of ESA treatment during cycles 1 to 8.
Time Frame: as for outcome 34
Population: as for outcome 40
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 97
percentage of participants | 30 (4.6) [15 to 45]

43. Secondary Outcome: Percentage of Participants Who Received ESAs and Achieved Hemoglobin From 10 to 12 g/dL 9 Weeks After Initiation of ESA Treatment
Description: The percentage of participants achieving a hemoglobin level from 10 to 12 g/dL after 9 weeks of ESA treatment.
Time Frame: 9 weeks post initiation of ESA treatment
Population: Participants who received treatment with an ESA
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 147
percentage of participants | 15 (4.6) [10 to 22]

44. Secondary Outcome: Number of Participants With Systemic Transfusions in Cycles 1 to 8
Description: Number of participants who received transfusions, including platelets, packed red blood cells, whole blood, or other, during cycles 1 to 8.
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 157 | 224 | 137 | 738 | 90 | 829
participants | 20 | 23 | 26 | 25 | 4 | 29

45. Secondary Outcome: Number of Transfusions Per Participant in Cycles 1 to 8
Time Frame: Cycles 1 - 8 (approximately 24 weeks)
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Number analyzed (Participants) | 157 | 224 | 137 | 738 | 90 | 829
participants
  No Transfusions | 137 | 201 | 111 | 713 | 86 | 800
  1 Transfusion | 8 | 16 | 17 | 19 | 2 | 21
  2 Transfusions | 4 | 4 | 5 | 3 | 1 | 4
  > 2 Transfusions | 8 | 3 | 4 | 3 | 1 | 4

ADVERSE EVENTS:
Time Frame: Approximately 24 weeks (8 treatment cycles)
Description: Only adverse drug reactions (ADRs) considered by the investigator to be related to Amgen products were collected. Any ADRs relating to pegfilgrastim, filgrastim, and darbepoetin alfa are reported.
  Other Adverse Events summarizes the non-serious occurrences of ADRs that exceed the 5% frequency threshold.
Groups:
- Ovarian: Ovarian Cancer
- NSCLC: Non-small Cell Lung Cancer
- SCLC: Small Cell Lung Cancer
- Breast Stage I-III: Breast Cancer, Stages I-III
- Breast Metastatic: Breast Cancer, Metastatic
- Breast Total: All Breast Cancer
Arm/Group | Ovarian | NSCLC | SCLC | Breast Stage I-III | Breast Metastatic | Breast Total
Serious Adverse Events (participants affected / at risk) | 0/157 | 1/224 | 0/137 | 1/738 | 0/90 | 1/829
Other Adverse Events (participants affected / at risk) | 1/157 | 0/224 | 1/137 | 37/738 | 1/90 | 38/829
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ovarian (N=157) | NSCLC (N=224) | SCLC (N=137) | Breast Stage I-III (N=738) | Breast Metastatic (N=90) | Breast Total (N=829)
CHEST PAIN (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ovarian (N=157) | NSCLC (N=224) | SCLC (N=137) | Breast Stage I-III (N=738) | Breast Metastatic (N=90) | Breast Total (N=829)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 37 | 1 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.